CLINICAL TRIAL: NCT05500742
Title: The proBNPage Reduction (PBAR) Randomized Trial: a Pilot Study to Define the Characteristics of Future Randomized Trials Aimed at Evaluating the Effects of Anti-aging Treatments on a Surrogate of Biological Age in Healthy Older Adults
Brief Title: Anti-age Dietary Supplements in Healthy Older Adults: the proBNPage Reduction Trial
Acronym: PBAR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Collaborators: University of Bologna (Other); Azienda Usl di Bologna (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PBAR-2022
Record Dates: First submitted 2022-08-09; First posted 2022-08-15 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2022-11

CONDITIONS: Aging
Keywords: Aging; Anti-age treatments; NT-proBNP; Coenzyme Q10; Selenium; Resveratrol; TA-65
MeSH Terms: interventions — coenzyme Q10; Selenium; Resveratrol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Coenzyme Q10 + Selenium (Active Comparator): Coenzyme Q10 100 mg bid + Selenium 100 mcg with the evening meal
  Interventions: Dietary Supplement: Coenzyme Q10; Dietary Supplement: Selenium
- Resveratrol + TA-65 (Active Comparator): Resveratrol 350 mg bid + TA-65 MD 100 U with the evening meal
  Interventions: Dietary Supplement: Resveratrol; Dietary Supplement: TA-65 MD
- Placebo (Placebo Comparator): Placebo-1 bid + Placebo-2 with the evening meal
  Interventions: Other: Placebo-1; Other: Placebo-2

INTERVENTIONS:
Dietary Supplement: Coenzyme Q10 — Soft 100 mg capsules containing coenzyme Q10 in vegetable oil provided by Pharma Nord
  Other Names: Q10 Gold
  Arms: Coenzyme Q10 + Selenium
Dietary Supplement: Selenium — 100 mcg tablets provided by Pharma Nord
  Other Names: SelenoPrecise
  Arms: Coenzyme Q10 + Selenium
Dietary Supplement: Resveratrol — 350 mg capsules provided by NOW Foods
  Other Names: Extra Strength Resveratrol
  Arms: Resveratrol + TA-65
Dietary Supplement: TA-65 MD — 100 unit capsules provided by TA Sciences
  Arms: Resveratrol + TA-65
Other: Placebo-1 — Soft capsules containing vegetable oil, externally identical to coenzyme Q10 capsules, provided by Pharma Nord
  Arms: Placebo
Other: Placebo-2 — Tablets containing excipients, externally identical to selenium tablets, provided by Pharma Nord
  Arms: Placebo

SUMMARY:
Background - The research on the possibilities to extend longevity in humans is presently based on large and long randomized longitudinal studies designed to compare all-cause mortality between treated and control groups. The availability of a simple and reliable marker of biological age might allow an acceleration of the research in this field, demonstrating in small samples and after limited periods of time, the ability of a given treatment to slow down, arrest or even revert the progression of biological age. Our previous studies suggest that this marker of biological age might be the N-terminal of B-type natriuretic peptide precursor (NT-proBNP), from which proBNPage, namely a biological age surrogate in years, can easily be calculated.

Objectives of the study - 1) To fine-tune the method of proBNPage assessment, i.e., to establish the minimum time required to detect a significant increase in proBNPage in a small group of subjects. This will be the duration of next studies to test possible "anti-age" treatments. 2) To assess the ability of 4 "anti-age" treatments, which provided promising results in previous experimental and human studies, to modify proBNPage progression.

Study design - Double-blind randomized clinical trial on a sample of healthy older adults stratified for age and sex.

Study description - One hundred and twenty healthy subjects (in particular, without previous or current cardiovascular diseases) aged 65-80 years of both sexes will be randomized into 3 groups: A) Coenzyme Q10 100 mg bid + Selenium 100 mcg; B) Resveratrol 350 mg bid + TA-65 MD 100 U; C) Placebo-1 bid + Placebo-2. All these subjects will be followed for 2 years and checked 8 times, to assess both proBNPage progression and the safety of the treatments. Handgrip strength, aerobic capacity at the step test and quality of life will also be assessed.

Statistical analysis - In the placebo group, the minimum time required to obtain a significant increase in proBNPage will be established by paired t tests. In the treated groups, possible differences in proBNPage progression with the curve obtained in the placebo group will be sought, both according to intention to treat and in the subjects that will complete the study, by repeated measures ANOVA.

DETAILED DESCRIPTION:
A) Background

Human life is relatively long so that, to assess the effect of any treatment on longevity, similarly long studies are needed. In addition, to demonstrate significant reductions in mortality, large samples are needed too. Thus, even though several promising treatments have been found in animal models, evidence of efficacy in humans has not come yet.

In an attempt to overcome these difficulties, several indicators of biological age have been proposed. Biological age may be defined as a measure, more reliable than chronological age, of how close to death an individual is. If such an indicator were available, assessing the efficacy of possible treatments would be relatively easy: one or two years of follow-up in relatively small groups might be sufficient to ascertain the arrest or even the inversion of the rise of the indicator.

In 2020 the authors proposed a new simple method to estimate a surrogate of biological age, the "proBNPage", starting from a single laboratory variable, NT-proBNP (the N-terminal fragment of type-B natriuretic peptide precursor). NT-proBNP is easily measurable in most laboratories. It is commonly used as a marker of heart failure, as it is released from the ventricular and atrial myocardium undergoing mechanical or ischemic stress. Several studies (both cross-sectional and longitudinal) have shown that this marker progressively increases with age. It is a good indicator of the risk of death even in subjects without cardiovascular diseases and, in particular, the authors have shown that NT-proBNP is associated with cardiovascular and all-cause mortality more strongly than chronological age. In addition, NT-proBNP is correlated with chronological age more strongly than all the main laboratory variables that had previously been proposed as biomarkers of biological age (as shown by the authors and subsequently also by others). Thus, starting from the equations of the regression lines of chronological age with NT-proBNP, the authors obtained two simple formulas, one for each sex, which allow the calculation of "proBNPage", in years, from the blood concentration of NT-proBNP.

Besides total and cardiovascular mortality, the authors have shown that other indicators of aging are independently associated with proBNPage, such as disease count, walking problems, the fitness assessed with a two-step test and the self-assessment of health status, in addition to previous myocardial infarction, previous stroke, peripheral artery disease and previous arterial revascularizations. Furthermore, in a recent study by other investigators, among more than 35000 clinical and laboratory biomarkers obtained from genomic, proteomic and metabolomic data in 4 cohorts of European populations, NT-proBNP was the marker most strongly associated with frailty in subjects without disability. Finally, in an older adult population, a further recent study has shown that NT-proBNP was the only independent risk factor of reduced intrinsic capacity among 20 laboratory variables, being associated with locomotion, hearing and vision disturbances and with some characteristic psychological aspects of aging.

To test, for the first time, the possible practical use of proBNPage, the authors have designed a study aimed at assessing the effects induced on it by a series of anti-age dietary supplements, which in previous studies have provided interesting results. For the choice of the treatments, the authors have sought the best compromise among available scientific evidence, safety and ease of obtaining the substances on the market.

Coenzyme Q10 (CoQ10): it is the only antioxidant that has been demonstrated to reduce cardiovascular mortality, in combination with selenium, in a sample of general population.

Selenium: selenoproteins contribute to the antioxidant systems of our organism. In addition, selenium has anti-inflammatory effects and is involved in the metabolism of thyroid hormones.

Resveratrol: powerful antioxidant, possible telomerase activator and inhibitor of the target of rapamycin (TOR) system.

TA-65: telomerase activator derived from Astragalus Membranaceus with proven capacity to lengthen telomeres in humans.

B) Study description

Design: Double-blind clinical trial with stratified randomization into 3 treatment groups (one placebo group and two food supplement-treated groups)

Primary objective: To describe, in the context of a longitudinal study lasting 2 years, the spontaneous trend of proBNPage in the placebo group, in order to find the parameters (time to reach a significant increase, magnitude of the increase and its variability) useful for planning future studies on anti-aging treatments.

Secondary objective: To describe, with pilot study, the potential of the proposed treatments to limit the progression of proBNPage, over the 2 years of study, compared to what is observed in the placebo group, to explore the feasibility and organizational needs of future multicenter trials on anti-aging treatments.

Study duration: 2 years

Sample size: 3 groups of 40 subjects each = 120 subjects

Non-institutionalized healthy elderly volunteers of both sexes will be included in the study. Their names and addresses will be obtained from lists provided by the public health service, including subjects aged 65-80 years, taking no more than 4 drugs a day and without recent (< 3 years) hospital admissions. By random choice, 2000 subjects with the above characteristics will receive a letter with the invitation to participate, together with a short questionnaire for preliminary health status assessment. For acceptation, the volunteers will return the compiled questionnaire by mail. Five hundred are expected to respond and, according to the information provided with the questionnaires, 200 of them will be selected (see inclusion and exclusion criteria) and summoned by phone for the first visit.

Screening assessment (Visit 1) After signing the informed consent, the subjects willing to participate will undergo anamnestic investigation (previous diseases, life habits, basal activities of daily living (ADL), instrumental activities of daily living (IADL), risk factors and medications taken, with all available documentation checked), medical examination (with weight, height, blood pressure and oxygen saturation), ECG and fasting venous blood sampling (for complete blood count, total cholesterol, HDL cholesterol, triglycerides, creatinine, Na, K, Ca, glutamic oxaloacetic transaminase, glutamic pyruvic transaminase, gamma glutamyl transpeptidase, creatine phosphokinase, erythrocyte sedimentation rate, C-reactive protein, blood glucose, glycated hemoglobin, international normalized ratio, activated partial thromboplastin time, and (in men) total and free prostate-specific antigen). According to the inclusion and exclusion criteria, 120 subjects will be selected to be randomized.

Randomization

The 120 selected patients will be subdivided into 4 strata with the following characteristics:

Men with age >= the median age of men

Men with age < the median age of men

Women with age >= the median age of women

Women with age < the median age of women

Using randomization lists, the subjects belonging to each stratum will be equally distributed among the 3 treatment groups, so that relevant casual displacements of age and sex among the groups will be avoided.

Baseline assessment (Visit 2) The selected subjects will undergo venous blood sampling for NT-proBNP measurement. This will be performed by fluorescence immune assay, using commercially available kits (Quidel).

Subsequent assessments: Visit 3: 14 days - Visit 4: 3 months - Visit 5: 6 months - Visit 6: 12 months - Visit 7: 18 months - Visit 8: 24 months.

Scheduled activities

Verification of safety of dietary supplements with: a) questionnaire for possible adverse reactions (all Visits); b) blood tests (like at Visit 1), ECG, body weight, blood pressure and oxygen saturation (Visits 1,3,4,6,8).

Longitudinal changes of proBNPage, with measurement of NT-proBNP (Visits 2,5,6,7,8).

Assessment of possible effects of dietary supplements on functional frailty indicators: a) Step test; b ) Handgrip; c) Euro QoL-5 Dimension questionnaire (Visits 2,5,6,7,8).

Every 6 months, handing of treatment boxes, collection of previous packages and check of treatments really taken (Visits 2,5,6,7,8).

Verification of possible adverse events, intervened diseases or variations of therapy and search for causes of possible deaths (all Visits)

C) Statistical analysis

Sample size was calculated with the goal of having, in repeated measures ANOVA, a probability of first type error < 0.05 and a probability of second type error < 0.20 (power 0.80). Using parameters obtained in our previous studies, the minimum size for each group was 9 (for between-within interaction). To account for probable dropouts, and to allow possible subgroup analysis, a fourfold sample will be opportune, that is, with 40 subjects per group.

Statistical procedures The primary objective of the study (establishing the time to reach a significant increase of proBNPage, the magnitude of the increase and its variability) requires the comparison, with Student's t for paired data, of proBNPage values at Visits 5 (6 months), 6 (12 months), 7 (18 months) and 8 (24 months) with the value at Visit 2 (baseline) in the placebo group.

The effects of treatments will be assessed considering both the completed cases and an intention-to-treat model. The variations (delta) of proBNPage within groups will be compared between groups by repeated measures ANOVA, with reference to the "between-within interaction". Two-tailed tests will be performed throughout, and P values < 0.05 will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

1. Age ranging between 65 and 80 years
2. Signed informed consent

Exclusion Criteria:

1. Previous or current atrial fibrillation
2. History of heart failure
3. History of coronary artery disease (myocardial infarction or angina pectoris)
4. Taking any of the dietary supplements of the present study during the 2 previous months
5. Taking a statin
6. Taking an anticoagulant drug
7. Taking more than 4 drugs a day
8. Hospital admission during the last 3 years
9. Known allergy to any drug of the present study
10. Malignant neoplasm in progress
11. Any other severe disease which, in the opinion of the investigator, contraindicates the participation in the study.
12. Alcohol or drug abuse
13. Participation in other trial
14. Uncertainty of the subject about his/her willingness to follow the study for 2 years
15. Deficit of one or more Activities of Daily Living (ADL)
16. Relevant alterations in the ECG or in the laboratory investigations which, in the opinion of the investigator, contraindicate the participation in the study.

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 120 (Actual)
Dates: Start 2022-07-22 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Change from baseline ProBNPage at 6 months | 6 months
  Change of surrogate, in years, of biological age, derived from mathematical transformation of NT-proBNP blood concentration with separate formulas for the two sexes
Change from baseline ProBNPage at 12 months | 12 months
  Change of surrogate, in years, of biological age, derived from mathematical transformation of NT-proBNP blood concentration with separate formulas for the two sexes
Change from baseline ProBNPage at 18 months | 18 months
  Change of surrogate, in years, of biological age, derived from mathematical transformation of NT-proBNP blood concentration with separate formulas for the two sexes
Change from baseline ProBNPage at 24 months | 24 months
  Change of surrogate, in years, of biological age, derived from mathematical transformation of NT-proBNP blood concentration with separate formulas for the two sexes

SECONDARY OUTCOMES:
Handgrip strength change | Baseline, 6 months, 12 months, 18 months, 24 months
  Strength of handgrip measured in Kg with dynamometer
Step test change | Baseline, 6 months, 12 months, 18 months, 24 months
  Time in seconds to ascend and descend 2 steps 20 times, inversely proportional to aerobic capacity
Euro QoL 5 dimension questionnaire change | Baseline, 6 months, 12 months, 18 months, 24 months
  Questionnaire including 5 questions on quality of life generating a synthetic score (EQ-5D Index) ranging from 0 (worst possible health status) to 1 (best possible health status)
Euro QoL 5 dimension Visual Analog Scale change | Baseline, 6 months, 12 months, 18 months, 24 months
  Visual Analog Scale (VAS) ranging from 0 (worst possible health status) to 100 (best possible health status)

CONTACTS AND LOCATIONS:
Overall Officials: Paola Forti, MD, Principal Investigator — University of Bologna and IRCCS Azienda Ospedaliero-Universitaria di Bologna, Italy
Locations (1):
- S. Orsola Hospital, Bologna, Italy

IPD SHARING:
Plan to Share IPD: Yes
All individual patient data that underlie results in a publication will be available to other researchers, upon reasonable request, after publication of study results.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available for 10 years after publication of study results
Access Criteria: Email request to principal investigator

REFERENCES:
- [Background] Muscari A, Bianchi G, Forti P, Magalotti D, Pandolfi P, Zoli M; Pianoro Study Group. N-terminal pro B-type natriuretic peptide (NT-proBNP): a possible surrogate of biological age in the elderly people. Geroscience. 2021 Apr;43(2):845-857. doi: 10.1007/s11357-020-00249-2. Epub 2020 Aug 11. PMID 32780292
- [Background] Muscari A, Bianchi G, Forti P, Giansante C, Giovagnoli M, Magalotti D, Pandolfi P, Perlangeli V, Zorzi V, Zoli M; Pianoro Study Group. A comparison of risk factors as predictors of cardiovascular and non-cardiovascular mortality in the elderly people--relevance of N-terminal pro-B-type natriuretic peptide and low systolic blood pressure. Int J Clin Pract. 2013 Nov;67(11):1182-91. doi: 10.1111/ijcp.12195. PMID 24165431
- [Background] Crimmins EM, Thyagarajan B, Kim JK, Weir D, Faul J. Quest for a summary measure of biological age: the health and retirement study. Geroscience. 2021 Feb;43(1):395-408. doi: 10.1007/s11357-021-00325-1. Epub 2021 Feb 5. PMID 33544281
- [Background] Muscari A, Bianchi G, Forti P, Magalotti D, Pandolfi P, Zoli M; Pianoro Study Group. The association of proBNPage with manifestations of age-related cardiovascular, physical, and psychological impairment in community-dwelling older adults. Geroscience. 2021 Aug;43(4):2087-2100. doi: 10.1007/s11357-021-00381-7. Epub 2021 May 13. PMID 33987773
- [Background] Gomez-Cabrero D, Walter S, Abugessaisa I, Minambres-Herraiz R, Palomares LB, Butcher L, Erusalimsky JD, Garcia-Garcia FJ, Carnicero J, Hardman TC, Mischak H, Zurbig P, Hackl M, Grillari J, Fiorillo E, Cucca F, Cesari M, Carrie I, Colpo M, Bandinelli S, Feart C, Peres K, Dartigues JF, Helmer C, Vina J, Olaso G, Garcia-Palmero I, Martinez JG, Jansen-Durr P, Grune T, Weber D, Lippi G, Bonaguri C, Sinclair AJ, Tegner J, Rodriguez-Manas L; FRAILOMIC initiative. A robust machine learning framework to identify signatures for frailty: a nested case-control study in four aging European cohorts. Geroscience. 2021 Jun;43(3):1317-1329. doi: 10.1007/s11357-021-00334-0. Epub 2021 Feb 18. PMID 33599920
- [Background] Ma L, Zhang Y, Liu P, Li S, Li Y, Ji T, Zhang L, Chhetri JK, Li Y. Plasma N-Terminal Pro-B-Type Natriuretic Peptide Is Associated with Intrinsic Capacity Decline in an Older Population. J Nutr Health Aging. 2021;25(2):271-277. doi: 10.1007/s12603-020-1468-3. PMID 33491044
- [Background] Alehagen U, Johansson P, Bjornstedt M, Rosen A, Dahlstrom U. Cardiovascular mortality and N-terminal-proBNP reduced after combined selenium and coenzyme Q10 supplementation: a 5-year prospective randomized double-blind placebo-controlled trial among elderly Swedish citizens. Int J Cardiol. 2013 Sep 1;167(5):1860-6. doi: 10.1016/j.ijcard.2012.04.156. Epub 2012 May 23. PMID 22626835
- [Background] Salvador L, Singaravelu G, Harley CB, Flom P, Suram A, Raffaele JM. A Natural Product Telomerase Activator Lengthens Telomeres in Humans: A Randomized, Double Blind, and Placebo Controlled Study. Rejuvenation Res. 2016 Dec;19(6):478-484. doi: 10.1089/rej.2015.1793. Epub 2016 Mar 30. PMID 26950204
- [Derived] Muscari A, Forti P, Brizi M, Magalotti D, Capelli E, Poti S, Piro F, Pandolfi P, Perlangeli V, Ramazzotti E, Barbara G; PBAR Study Group. Can We Slow Down Biological Age Progression? Study Protocol for the proBNPage Reduction (PBAR) Randomized, Double-Blind, Placebo-Controlled Trial (Effects of 4 "Anti-Aging" Food Supplements in Healthy Older Adults). Clin Interv Aging. 2023 Oct 27;18:1813-1825. doi: 10.2147/CIA.S422371. eCollection 2023. PMID 37915546